CLINICAL TRIAL: NCT03028389
Title: Effects of Limb Remote Ischemic Preconditioning for Prevention of Delirium in Elderly Patients After Non-cardiac Surgery:a Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Effects of Limb Remote Ischemic Preconditioning for Prevention of Delirium in Elderly Patients After Non-cardiac Surgery
Acronym: LRIP-D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Kexuan Liu, Department of Anesthesiology, Nanfang Hospital, Southern Medical University, Guangzhou, China, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LRIP20170116
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Elderly Patients; Non-cardiac Surgery
Keywords: elderly patients; non-cardiac surgery; ischemic preconditioning; delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Limb RIPC (Experimental): The limb RIPC protocol was applied after anesthetic induction and before the start of surgery. The limb RIPC was induced by placing a blood pressure cuff on the left upper arm of patient for three inflating-deflating cycles: 5 min inflating to 200 mmHg followed by a 5 min reperfusion with deflating the cuff.
  Interventions: Procedure: limb remote ischemic preconditioning(LRIP)
- Convention (No Intervention): Elderly patients undergoing non-cardiac surgery received no treatment after induction of anaesthesia

INTERVENTIONS:
Procedure: limb remote ischemic preconditioning(LRIP) — LRIP consisted of three cycles of left upper limb ischemia induced by inflating a blood pressure cuff on the left upper arm to 200mmHg, with an intervening 5 minutes of reperfusion, during which time the cuff was deflated.
  Other Names: LRIP
  Arms: Limb RIPC

SUMMARY:
To investigate whether limb remote ischemic preconditioning (LRIP) could safely decrease the incidence of delirium in elderly patients after non-cardiac surgery.

DETAILED DESCRIPTION:
Remote ischaemic preconditioning may confer the cytoprotection in critical organs. We hypothesized that limb remote ischemic preconditioning (RIPC) would safely decrease the incidence of delirium in elderly patients after non-cardiac surgery.The primary outcomes included the incidence of delirium in the first 7 days after surgery using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) scale.The quality of recovery over a 6-month period was evaluated as well.Secondary endpoints included length of stay in the hospital after surgery (from day of surgery to hospital discharge), occurrence of non-delirium postoperative complications, and all-cause 6-month mortality.

ELIGIBILITY:
Inclusion Criteria:

* elderly patients received elective non-cardiac surgery with general anesthesia
* anticipated surgery time > 2 hours

Exclusion Criteria:

* age < 65 years old
* Acute coronary syndrome or myocardial infraction within 3 months
* Chronic obstructive pulmonary emphysema
* Serious hepatic dysfunction (Child-Pugh class C)
* serious renal dysfunction (undergoing dialysis before surgery)
* Ejection fraction less than 40%
* Poor pulmonary function (PaO2 <60mmHg)
* Preoperative history of schizophrenia, epilepsy, Parkinsonism, or myasthenia gravis
* Inability to communicate in the preoperative period (coma, profound dementia, or language barrier)
* Brain injury or neurosurgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 611 (Estimated)
Dates: Start 2017-02-01 (Estimated); Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
the incidence of delirium | in the first 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Xuan Liu, Ph.D, Principal Investigator — Nanfang Hospital, the Southern Medical University

IPD SHARING:
Plan to Share IPD: No